CLINICAL TRIAL: NCT02451969
Title: Phase III Safety and Immunogenicity Study of 23-valent Pneumococcal Polysaccharide Vaccine: A Double-blind, Randomized and Controlled Clinical Trial With 23-valent Pneumococcal Polysaccharide Vaccine in Healthy Children, Adults, and Elderly
Brief Title: Safety and Immunogenicity Study of 23-valent Pneumococcal Polysaccharide Vaccine in Healthy Children, Adults and Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PPV-3001
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2015-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0
  * Intervention: investigational 23-valent PPV
  Interventions: Biological: investigational 23-valent PPV
- Control Group (Active Comparator): * Single intramuscular injection of the control vaccine (0.5 ml) on Day 0
  * Intervention: control 23-valent PPV
  Interventions: Biological: control 23-valent PPV

INTERVENTIONS:
Biological: investigational 23-valent PPV — The investigational vaccine was manufactured by Sinovac Biotech Co., Ltd.
  Arms: Experimental Group
Biological: control 23-valent PPV — The control vaccine was manufactured by Chengdu Institute of Biological products Co., Ltd.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of an investigational 23-valent pneumococcal polysaccharide vaccine (PPV) in healthy children, adults and elderly. The control vaccine is a commercialized 23-valent PPV.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, single-center, controlled phase III clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of an investigational 23-valent pneumococcal polysaccharide vaccine (PPV) manufactured by Sinovac Biotech Co., Ltd. The primary objective of this study is to demonstrate that the immunogenicity of the investigational vaccine is non-inferior to that of a commercialized 23-valent PPV manufactured by Chengdu Institute of Biological products Co., Ltd.; the secondary objective is to assess the safety of the investigational and control vaccines. Participants will be grouped into three cohorts by age: child cohort (2 - 17 years old), adult cohort (18 - 60 years old) and elderly cohort (≥ 61 years old). In each cohort, the participants will be randomly assigned into experimental group or control group in the ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer ≥ 2 years old;
* Proven legal identity;
* Written consent of the guardian of participants < 18 years old, and written consent of the participant ≥ 12 years old;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* Prior vaccination with pneumococcal vaccine;
* History of bacterial pneumonia within 3 years prior to this study;
* Pregnant, breast feeding, or women expected to conceive within 60 days after vaccination;
* History of allergy to any vaccine or vaccine ingredient;
* Receipt of any of the following products:

  1. Blood product within 3 months prior to study entry;
  2. Any live attenuated vaccine within 28 days prior to study entry;
  3. Any subunit vaccine or inactivated vaccine within 14 days prior to study entry;
  4. Any immunosuppressant within 6 month prior to study entry;
* Congenital malformation, developmental disorders, serious chronic diseases, autoimmune disease, immunodeficiency, serious cardiovascular disease, diabetes, hypertension that cannot be stabilized by medication, liver or kidney disease, or malignant tumor;
* History of asthma, thyroidectomy, angioneurotic edema, severe nervous system disease or mental illness; without spleen or splenectomy; diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities), or obvious bruising or coagulation disorders;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillaty temperature > 37.0 °C;
* Any other factor that in the opinion of the investigator suggesting the volunteer is unsuitable for this study;
* Participants with the following conditions from day 0 - 28 would be included in the full analysis set (FAS), but would be excluded from the per protocol set (PPS):

  1. Receipt of any other investigational or unregistered product (drug or vaccine);
  2. Receipt of immunosuppressant (corticosteroid dosage that equivalent to or above 0.5 mg prednisone/kg weight/day) for > 14 days, except for inhalant or locally administrated corticosteroid;
  3. Receipt of immunoglobulin and/or blood product;
  4. Newly diagnosed autoimmune disease or immunodeficiency (e.g., HIV infection);

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1760 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCR) of each of the 23 pneumococcal serotypes | 28 days
  For each serotype, the SCR is the percentage of participants with the increase of relative antibody concentration ≥ 2 folds after vaccination. The relative antibody concentrations were measured using Enzyme Linked Immunosorbent Assay (ELISA).

SECONDARY OUTCOMES:
The incidences of adverse events (AEs) | 28 days
  After each injection, a 30-minute safety observation was conducted immediately. The body temperature, occurrence of solicited local and general AEs on day 0 - 7 were reported. Unsolicited AEs occurred during day 0 - 28 were also reported. Each AE case was reviewed by the investigator to determine whether or not it was an adverse reaction (related to the vaccination).
The increases of relative antibody concentration against each of the 23 pneumococcal serotypes | 28 days
  The relative antibody concentrations in the pre- and post-immunization serum samples were measured using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Ru, BS, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Kaifeng County Center for Disease Control and Prevention, Kaifeng, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang L, Wang L, Li H, Hu Y, Ru W, Han W, Shi G, Ye Q, Han Z, Xia J, Xia S, Xu M, Li J. A phase III clinical trial to evaluate the safety and immunogenicity of 23-valent pneumococcal polysaccharide vaccine (PPV23) in healthy children, adults, and elderly. Hum Vaccin Immunother. 2019;15(1):249-255. doi: 10.1080/21645515.2018.1509648. Epub 2018 Sep 21. PMID 30215583